CLINICAL TRIAL: NCT04187417
Title: Short Term Topical Tetracaine is Safe and Highly Efficacious for the Treatment of Pain Caused by Corneal Abrasions: a Double-blind Randomized Clinical Trial
Brief Title: Short Term Topical Tetracaine is Safe and Highly Efficacious for the Treatment of Pain Caused by Corneal Abrasions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: INTEGRIS Southwest Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-055
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Corneal Abrasion
MeSH Terms: conditions — Corneal Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: sealed, numbered opaque envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical tetracaine (Experimental): Topical tetracaine hydrochoride 1%
  Interventions: Drug: topical tetracaine hydrochloride 1%
- Balanced artificial tear solution (Placebo Comparator): Balanced artificial tear solution (Systane)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: topical tetracaine hydrochloride 1% — topical ophthalmologic anesthestic
  Arms: Topical tetracaine
Drug: Placebo — Placebo
  Arms: Balanced artificial tear solution

SUMMARY:
The objective of this study was to show that patients with corneal abrasions would experience more pain relief with short term topical tetracaine than placebo, have similar complication rates, and take less hydrocodone for breakthrough pain.

DETAILED DESCRIPTION:
Corneal abrasions are among the most common eye-related injuries seen in the emergency department (ED). Topical anesthetic drops are routinely used prior to slit-lamp examination for diagnosis of corneal abrasions and often provide immediate pain relief. Patients are then sent home with oral analgesics and topical antibiotics. The use of topical anesthetics for outpatient treatment of corneal abrasions is discouraged by most emergency medicine textbooks due to concerns over safety. Case reports of abuse and misuse as well as animal studies have suggested that long term use of topical anesthetics may lead to rare complications. Two clinical trials showed no delayed healing after a short course of topical anesthetics following PRK surgery. Whether this could be applied to nonsurgical patients in the ED was investigated by two small clinical trials that showed similar efficacy and safety but were underpowered to prove a statistical difference. In 2014, a larger randomized trial demonstrated the safety of tetracaine for ED patients with corneal abrasions but failed to show a significant difference in patient visual analogue scale (VAS) pain ratings over time. More recently, a retrospective cohort study of 444 ED patients given tetracaine for 24 hours reported no serious complications or uncommon adverse events. If topical anesthetics could be safely prescribed for short term use in the management of corneal abrasions, it is possible that this would decrease use of systemic opioids for this purpose. The aim of this randomized, double-blind trial was to compare the effectiveness of topical tetracaine versus placebo in ED patients with corneal abrasions as measured by a reduction in the VAS score.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years to 80 years old presenting to the ED with suspected acute corneal abrasion from mechanical trauma or removal of a foreign body by the physician were included

Exclusion Criteria:

* Patients were excluded if they wore contact lenses, had previous corneal surgery or transplant in the affected eye, presented more than 36 hours after their injury, had a grossly contaminated foreign body or coexisting ocular infection. Additional exclusion criteria were pregnancy, retained foreign body, penetrating eye injury, immunosuppression, allergy to study medication, inability to attend follow up, inability to fluently read and speak English or Spanish, or any injury requiring urgent ophthalmologic evaluation (large or complicated abrasions with significant vision loss, corneal ulcers, corneal lacerations).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Overall Visual Analog Scale score | 48 hours
  The primary endpoint of the study was the overall post study drop Visual Analog Scale pain score measured at the patients initial follow up Emergency Department visit. Measured on a 0-10 scale with 0 meaning no pain and 10 worst pain.

SECONDARY OUTCOMES:
Visual Analog Scale score | 1 week
  Secondary endpoint were the average self-reported post study drop Visual Analog Scale score after each use.Measured on a 0-10 scale with 0 meaning no pain and 10 worst pain.
Number of hydrocodone tablets taken | 48 hours
adverse events | 1 week
  any adverse events

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waldman N, Winrow B, Densie I, Gray A, McMaster S, Giddings G, Meanley J. An Observational Study to Determine Whether Routinely Sending Patients Home With a 24-Hour Supply of Topical Tetracaine From the Emergency Department for Simple Corneal Abrasion Pain Is Potentially Safe. Ann Emerg Med. 2018 Jun;71(6):767-778. doi: 10.1016/j.annemergmed.2017.02.016. Epub 2017 May 5. PMID 28483289
- [Background] Waldman N, Densie IK, Herbison P. Topical tetracaine used for 24 hours is safe and rated highly effective by patients for the treatment of pain caused by corneal abrasions: a double-blind, randomized clinical trial. Acad Emerg Med. 2014 Apr;21(4):374-82. doi: 10.1111/acem.12346. PMID 24730399
- [Background] Ball IM, Seabrook J, Desai N, Allen L, Anderson S. Dilute proparacaine for the management of acute corneal injuries in the emergency department. CJEM. 2010 Sep;12(5):389-96. doi: 10.1017/s1481803500012537. PMID 20880433
- [Background] Ting JY, Barns KJ, Holmes JL. Management of Ocular Trauma in Emergency (MOTE) Trial: A pilot randomized double-blinded trial comparing topical amethocaine with saline in the outpatient management of corneal trauma. J Emerg Trauma Shock. 2009 Jan;2(1):10-4. doi: 10.4103/0974-2700.44676. PMID 19561949
- [Background] Verma S, Corbett MC, Patmore A, Heacock G, Marshall J. A comparative study of the duration and efficacy of tetracaine 1% and bupivacaine 0.75% in controlling pain following photorefractive keratectomy (PRK). Eur J Ophthalmol. 1997 Oct-Dec;7(4):327-33. doi: 10.1177/112067219700700404. PMID 9457454
- [Background] Verma S, Corbett MC, Marshall J. A prospective, randomized, double-masked trial to evaluate the role of topical anesthetics in controlling pain after photorefractive keratectomy. Ophthalmology. 1995 Dec;102(12):1918-24. doi: 10.1016/s0161-6420(95)30775-0. PMID 9098296
- [Background] Chang YS, Tseng SY, Tseng SH, Wu CL. Cytotoxicity of lidocaine or bupivacaine on corneal endothelial cells in a rabbit model. Cornea. 2006 Jun;25(5):590-6. doi: 10.1097/01.ico.0000220775.93852.02. PMID 16783149
- [Background] Grant RL, Acosta D. Comparative toxicity of tetracaine, proparacaine and cocaine evaluated with primary cultures of rabbit corneal epithelial cells. Exp Eye Res. 1994 Apr;58(4):469-78. doi: 10.1006/exer.1994.1040. PMID 7925683
- [Background] Bisla K, Tanelian DL. Concentration-dependent effects of lidocaine on corneal epithelial wound healing. Invest Ophthalmol Vis Sci. 1992 Oct;33(11):3029-33. PMID 1399407
- [Background] Higbee RG, Hazlett LD. Topical ocular anesthetics affect epithelial cytoskeletal proteins of wounded cornea. J Ocul Pharmacol. 1989 Fall;5(3):241-53. doi: 10.1089/jop.1989.5.241. PMID 2625618
- [Background] Rosenwasser GO, Holland S, Pflugfelder SC, Lugo M, Heidemann DG, Culbertson WW, Kattan H. Topical anesthetic abuse. Ophthalmology. 1990 Aug;97(8):967-72. doi: 10.1016/s0161-6420(90)32458-2. PMID 2402423
- [Background] Rosenwasser GO. Complications of topical ocular anesthetics. Int Ophthalmol Clin. 1989 Fall;29(3):153-8. doi: 10.1097/00004397-198902930-00005. No abstract available. PMID 2666331
- [Background] Henkes HE, Waubke TN. Keratitis from abuse of corneal anaesthetics. Br J Ophthalmol. 1978 Jan;62(1):62-5. doi: 10.1136/bjo.62.1.62. PMID 629912
- [Background] Willis WE, Laibson PR. Corneal complications of topical anesthetic abuse. Can J Ophthalmol. 1970 Jul;5(3):239-43. No abstract available. PMID 5472832
- [Background] Ahmed F, House RJ, Feldman BH. Corneal Abrasions and Corneal Foreign Bodies. Prim Care. 2015 Sep;42(3):363-75. doi: 10.1016/j.pop.2015.05.004. Epub 2015 Jul 31. PMID 26319343
- [Derived] Shipman S, Painter K, Keuchel M, Bogie C. Short-Term Topical Tetracaine Is Highly Efficacious for the Treatment of Pain Caused by Corneal Abrasions: A Double-Blind, Randomized Clinical Trial. Ann Emerg Med. 2021 Mar;77(3):338-344. doi: 10.1016/j.annemergmed.2020.08.036. Epub 2020 Oct 27. PMID 33121832